CLINICAL TRIAL: NCT04731012
Title: Immunological and Cardiovascular Phenotyping of Oocyte-donation Pregnancies
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Florian Herse, Doctor of Science, Charite University, Berlin, Germany
Other Study IDs: ED-S
Record Dates: First submitted 2020-09-21; First posted 2021-01-29 (Actual); Last update posted 2021-01-29 (Actual); Status verified 2021-01

CONDITIONS: Preeclampsia; Oocyte-donation Pregnancies
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- healthy oocyte-donation pregnancy: healthy pregnancy
- preeclamptic oocyte-donation pregnancy: preeclampsia
- healthy IVF or ICSI pregnancy: healthy pregnancy
- preeclamptic IVF or ICSI pregnancy: preeclampsia
- healthy spontaneous conception pregnancy: healthy pregnancy
- preeclamptic spontaneous conception pregnancy: preeclampsia

SUMMARY:
The investigators conduct a study to evaluate the underlying causes of preeclampsia in oocyte-donation pregnancies.

DETAILED DESCRIPTION:
A detailed medical history, questionnaires as well as blood, urine and placental samples will be used to analyse several factors leading to the high risk of preeclampsia in oocyte-donation pregnancies.

ELIGIBILITY:
Inclusion Criteria:

* pregnancy

Exclusion Criteria:

* severe auto immune disorders

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: * oocyte donation pregnancies
  * IVF or ICSI pregnanies
  * spontaneous conception pregnancies
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Preeclampsia in oocyte-donation pregnancies is caused by an altered composition of immune cells in placenta and blood. | 01.01.2020 - 01.12.2025
  T-Cell populations are altered in preeclampsia. HLA-mismatch of mother and donor oocyte lead to a "host-versus-graft" reaction. T-, B- and Natural killer cells are altered in placental tissue of oocyte-donation pregnancies.

SECONDARY OUTCOMES:
Preeclampsia in oocyte-donation pregnancies is caused by an activation of pro-inflammatory factors and endothelial dysfunction. | 01.01.2020 - 01.12.2025
  Altered Natural killer cells and B-cells in oocyte-donation pregnancies lead to endothelial dysfunction. Pro-inflammatory factors are higher in OD pregnancy and can be measured in placental tissue via single-cell sequencing.

CONTACTS AND LOCATIONS:
Locations (1):
- Experimental and Clinical Research Center (ECRC), Berlin, Germany

IPD SHARING:
Plan to Share IPD: Undecided